CLINICAL TRIAL: NCT06533163
Title: Low-Intensity Oscillatory Magnetic Therapy in Patients With Newly Diagnosed Glioblastoma Multiforme (GBM) - An Exposure-time Escalation Pilot Trial
Acronym: OMX-EFS-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: BioTex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMX-EFS-01
Record Dates: First submitted 2024-05-15; First posted 2024-08-01 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma Multiforme
MeSH Terms: conditions — Glioblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Device use (Experimental): This investigation will employ an individualized dose-time-escalation approach starting each patient at a low dose and escalating the dose within the same patient.
  For each patient, the device will be used starting at 4 hours per day. If a patient doesn't experience any issues for 2 weeks, they would ramp up to 6 hours per day. After another 2 weeks without issues, they will increase to 8 hours per day and maintain that for the remainder of the study.
  If a patient encounters any issues thought to probably be device related by the PI during any of the 2-week intervals at different doses, they will be reduced by 4 hours per day (with a minimum therapy of 2 hours per day) for a specified duration up to 2 weeks, although this can be adjusted based on symptoms at the investigator's discretion. Each patient will follow this personalized escalation pathway.
  Interventions: Device: Oncomagnetic device

INTERVENTIONS:
Device: Oncomagnetic device — OncoMAGNETX has developed a portable wearable noninvasive magnetic device (Oncomagnetic device) for the treatment of GBM.

SUMMARY:
The clinical investigation is a non-randomized, multicenter, open-label, prospective, exposure-time escalation clinical investigation. The clinical investigation is designed to assess the clinical safety and performance of the Oncomagnetic Device.

ELIGIBILITY:
Inclusion Criteria:

1. The subject is at least 18 years of age.
2. The subject previously had maximal safe resection (MSR) for glioblastoma (GBM) per the discretion of the investigator and is able to receive standard radiotherapy (unless contraindicated or refused by the subject)
3. The subject has a newly confirmed diagnosis of GBM per WHO classification criteria.
4. The subject has pre-op, post-surgical MRI and RX planning MRI scans available for Investigator review.
5. The subject has a confirmed unmethylated MGMT promoter status.
6. The subject has a KPS ≥ 70.
7. The subject's life expectancy is >12 weeks.
8. The subject is no longer taking corticosteroids.
9. The subject has signed and dated the consent form.
10. The subject has stated understanding and willingness to comply with all clinical investigation procedures and availability for the duration of the clinical investigation.

Exclusion Criteria:

1. The subject has a tumor in the brainstem, extensive or multicentric disease (e.g. in both hemispheres), or an abnormal regrowth pattern between the post operation MRI and RX planning MRI, suggesting early tumor progression, as determined by the Investigator's discretion.
2. The subject is any of the following: pregnant, planning on becoming pregnant during the investigation, breastfeeding, incarcerated, or enrolled in another clinical investigation.
3. The subject has a severe acute infection, any autoimmune disease, significant congenital anomaly, other co-morbidity, or medical problem or is taking immunosuppressant therapy (except Dexamethasone) within 90 days of anticipated device use for a condition that in the opinion of the Investigator and Sponsor precludes enrollment in the investigation.
4. The subject has had a known focal or generalized seizure after surgery.
5. The subject has implants or any condition preventing the patient from undergoing serial MRI scans.
6. The patient has a skull defect (such as, missing bone with no replacement), bullet fragments or ferrous metals.
7. The subject has an active implanted device (e.g., cardiac pacemakers, Vagus Nerve Stimulation [VNS], Deep Brain Stimulation [DBS], programmable shunts, etc.).
8. The subject has any of the following lab results:

   * ANC < 1000 cells/mm3 or < 1.5 x 10^9 /L.
   * Platelet count < 100,000 cells/mm3.
9. The subject has a history of any previous anti-tumor treatment for a brain tumor.
10. The subject is currently being treated or has been treated with other investigational agents/devices that may compromise the results of this investigation (as per discretion of the Investigator).
11. The subject takes any nutritional supplements or alternative medical treatments that may compromise the results of this investigation (this is as per discretion of the Investigator, but any compound with anti-oxidant properties is strongly discouraged).
12. The subject has planned concomitant or adjuvant chemotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-17 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
To assess the safety of the Oncomagnetic device. | 6 months
  • Incidence of device-related adverse events (as per CTCAE v.5) at 6 months following surgery.

SECONDARY OUTCOMES:
To evaluate the performance of the Oncomagnetic Device in patients with newly diagnosed GBM. | 6 months
  Response of Index Lesion:
  • Via radiographic assessment (MRI)
To evaluate the performance of the Oncomagnetic Device in patients with newly diagnosed GBM. | 6 months
  Median Progression-Free Survival at 6 months (PFS-6) following surgery:
  • Changes in tumor volume via radiographic assessment (MRI) analyzed via independent reviewer using mRANO criteria.
To evaluate the performance of the Oncomagnetic Device in patients with newly diagnosed GBM. | 3 years
  Median Overall Survival (OS):
  • Measured by the length of time from initial diagnosis until subject expiration.
To evaluate the performance of the Oncomagnetic Device in patients with newly diagnosed GBM. | 6 months
  Quality of Life (QOL):
  • Assessed using the validated quality of life scale (QLQ-C30) by the EORTC as well as the module for brain tumors, BN 20 and Barthel Index.

OTHER OUTCOMES:
To assess imaging data for exploratory analyses and to support potential future research endeavors. | 3 years
  • Via radiographic assessment (MRI)
To identify biomarkers that correlate with outcome. | 3 years
  Via blood biomarker collection

CONTACTS AND LOCATIONS:
Overall Officials: Frank Giordano, MD, Principal Investigator — Universitätsmedizin Mannheim | UMM
Locations (6):
- Germany (6):
  - Clinical Center Stuttgart, Stuttgart, Baden-Wurttemberg
  - Technical University of Munich, München, Bavaria
  - University Hospital Bonn, Bonn, North Rhine-Westphalia
  - Clinical Center Lünen, Lünen, North Rhine-Westphalia
  - University Hospital Leipzig, Leipzig, Saxony
  - Medical Center Mannheim, Mannheim

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared via Clinical Trial Journal
Supporting Information: CSR
Time Frame: After Study Completion